CLINICAL TRIAL: NCT03709355
Title: Open-Label Pharmacokinetics Study to Evaluate Drug-Drug Interactions and Safety of ELPIDA® in Co-Administration With Other Drugs in Healthy Volunteers
Brief Title: Pharmacokinetics Study to Evaluate Drug-Drug Interactions and Safety of Elpida® in Co-Administration With Other Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HIV-VM1500-08
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: HIV-1-infection
Keywords: HIV-1
MeSH Terms: interventions — elsulfavirine; Rifampin; Rifabutin; Clarithromycin; Omeprazole; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Elpida® single dose (Active Comparator): Single dose of Elpida® (capsule 20 mg)
  Interventions: Drug: Elpida®
- Rifampin & Elpida® (Experimental): Single dose of Rifampin (capsule 150 mg), Rifampin + Elpida® 20mg single dose
  Interventions: Drug: Elpida®; Drug: Rifampin
- Rifabutin & Elpida® (Experimental): Single dose of Rifabutin capsule 150 mg, Rifabutin + Elpida® 20mg single dose
  Interventions: Drug: Elpida®; Drug: Rifabutin
- Clarithromycin & Elpida® (Experimental): Single dose of Clarithromycin capsule 250 mg, Clarithromycin + Elpida® 20mg single dose
  Interventions: Drug: Elpida®; Drug: Clarithromycin
- Omeprazole & Elpida® (Experimental): Single dose of Omeprazole capsule 20 mg, Omeprazole + Elpida® 20mg single dose
  Interventions: Drug: Elpida®; Drug: Omeprazole
- Atorvastatin & Elpida® (Experimental): Single dose of Atorvastatin tablet 80 mg, Atorvastatin + Elpida® 20mg single dose
  Interventions: Drug: Elpida®; Drug: Atorvastatin
- Levonorgestrel+Ethinylestradiol & Elpida® (Experimental): Single dose of Levonorgestrel 150 µg + Ethinylestradiol 150 µg tablet, Levonorgestrel + Ethinylestradiol + Elpida® 20mg single dose
  Interventions: Drug: Elpida®; Drug: Levonorgestrel+Ethinylestradiol
- Elpida® multiple dose (Active Comparator): Elpida® QD dosing for 14 days
  Interventions: Drug: Elpida®

INTERVENTIONS:
Drug: Elpida® — Elpida® capsules, 20mg
  Other Names: elsulfavirine; VM1500; VM-1500
Drug: Rifampin — Rifampin capsules, 150mg
  Arms: Rifampin & Elpida®
Drug: Rifabutin — Rifabutin capsules, 150mg
  Arms: Rifabutin & Elpida®
Drug: Clarithromycin — Clarithromycin Film-coated tablets, 250mg
  Arms: Clarithromycin & Elpida®
Drug: Omeprazole — Omeprazole Film-coated tablets 20mg
  Arms: Omeprazole & Elpida®
Drug: Atorvastatin — Atorvastatin Film-coated tablets, 80mg
  Arms: Atorvastatin & Elpida®
Drug: Levonorgestrel+Ethinylestradiol — Levonorgestrel 150 μg + Ethinylestradiol 30 μg, Film-coated tablets
  Arms: Levonorgestrel+Ethinylestradiol & Elpida®

SUMMARY:
The study assesses PK and safety of other drugs, such as some antibiotics, proton pump inhibitors, statins, and combined oral contraceptives when co-administered with Elpida®

DETAILED DESCRIPTION:
This study evaluates the drug-drug interaction of Elpida® and other drugs (Rifampin, Rifabutin, Clarithromycin, Omeprazole, Atorvastatin and combinations of Levonorgestrel and Ethinylestradiol) according to changes in the PK parameters of the study substances in their single co-administration in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects must meet the following criteria to be enrolled in the study:

1. Non-smoking men and women between the ages of 18 and 45 years (inclusive) (only women in Group 7);
2. Verified "healthy" diagnosis according to standard clinical, laboratory and instrumental examination methods;
3. Body Mass Index ranges between 18.5 kg/m2 and 30.0 kg/m2 and a body weight NLT 50 kg;
4. Negative alcohol and drug tests;
5. Consent to use two adequate and reliable methods of contraception throughout the study and up to 3 months after its completion: a condom with spermicide (foam, gel, cream, suppositories), or a diaphragm with spermicide, or a condom and diaphragm, or a condom and an intrauterine device;
6. Signed Patient Information Sheet and form of Informed Consent to participate in the study.

Exclusion Criteria:

A subject will be considered not eligible to participate in the study if one or more of the following criteria is met:

1. Chronic diseases of cardiovascular, bronchopulmonary, neuroendocrine, musculoskeletal system, as well as diseases of the gastrointestinal tract, liver, kidneys, blood;
2. Variables of standard laboratory and instrumental parameters are beyond the normal limits (taking into account the acceptable limits of laboratory parameters;
3. Surgical interventions on the gastrointestinal tract in medical history (except appendectomy);
4. Systolic pressure below 90 mm Mercury or above 130 mm Mercury, diastolic pressure below 60 mm Mercury or above 85 mm Mercury, heart rate less than 60 BPM or more than 90 BPM at screening;
5. Regular intake of drugs less than 2 weeks prior to screening (including herbal preparations and dietary supplements); intake of drugs that have a pronounced effect on hemodynamics, hepatic function, etc. (for example, barbiturates, omeprazole, cimetidine, etc.) less than 30 days prior to screening;
6. Presence of antibodies to HIV and hepatitis C virus, presence of hepatitis В surface antigen, a positive syphilis test;
7. An unstable sleep structure (e.g., night work, sleep disorders, insomnia, recent return from another time zone, etc.), extreme physical activity (e.g. weight lifting), a special diet (e.g. vegetarian, vegan);
8. Signs of alcohol (intake of more than 10 units of alcohol per week) or drug addiction; alcohol or drugs consumption within 4 days prior to screening; cigarettes smoking 3 months prior to screening; positive drug and/or alcohol test;
9. Drug allergies in medical history (including drug intolerance, including hypersensitivity to any components of study drugs) as well as food allergy;
10. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption;
11. Individual intolerance to any components of study drugs;
12. Blood/plasma donation (450 ml of blood or plasma and more) less than 2 months prior to screening;
13. Treatment with a study drug in framework of other clinical trials within 1 month prior to screening (including follow-up visits);
14. Acute infectious diseases less than 4 weeks prior to screening;
15. Inhibitors or inducers of CYP3A4/5, drugs that cause QT prolongation within 30 days prior to StD administration;
16. For women - positive result of pregnancy test or breastfeeding; Inability to read or write; unwillingness to understand and adhere to the study protocol procedures; non-compliance with the drugs intake regimen or execution of procedures, which as the Investigator believes may affect the study results or subject's safety and prevent the subject from further participation in the study; any other associated medical or serious psychological conditions making the subject not eligible to participate in the clinical study, restricting legality of obtaining the Informed Consent or affecting the subject's ability to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of elsulfavirine | 42 days
Plasma concentration of VM1500A | 42 days
Plasma concentration of rifampicin | 42 days
Plasma concentration of rifabutin | 49 days
Plasma concentration of clarithromycin | 42 days
Plasma concentration of atorvastatin | 42 days
Plasma concentration of levonorgestrel | 42 days
Plasma concentration of ethinylestradiol | 42 days

SECONDARY OUTCOMES:
The incidence of AEs and SAEs | 49 days

CONTACTS AND LOCATIONS:
Overall Officials: Elena Smolyarchuk, PhD, Principal Investigator — I.M. Sechenov First Medical State University; Alla Andreeva, PhD, Principal Investigator — Smolensk Region Clinical Hospital
Locations (1):
- Central Clinical City Hospital, Reutov, Moscow Oblast, Russia